CLINICAL TRIAL: NCT04238494
Title: Muscle Multi-parametric NMR Imaging Development in Aged People With Sarcopenia or Frailty Syndrome; CLINical Study
Acronym: MIDAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2019/09
Record Dates: First submitted 2019-08-19; First posted 2020-01-23 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Frail Elderly Syndrome; Diabetes
Keywords: imaging; myosteatosis (Myosteatosis is the pathologic accumulation of lipid that can occur in conjunction with atrophy and fibrosis following skeletal muscle injury)
MeSH Terms: conditions — Diabetes Mellitus | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Multicomponent assessment: clinical, biological, functional, cognitive and MRI (muscle and brain)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Frail/prefrail (Experimental): Fried's criteria >3 = frail, 1 or 2 = prefrail The 5 Fried criteria mainly target the muscle function: low muscle strength, decreased physical activity and low gait speed. One refers to depressive symptoms with the use of 2 CES-D (Centre for Epidemiologic Studies - Depression Scale) questions and one to nutrition with the weight loss criteria. The second most famous definition of frailty was developed by ROCKWOOD and MITNISIKI (2). It describes frailty as the accumulation of deficits including cognitive, functional and social alterations
  Interventions: Diagnostic Test: Nuclear magnetic resonance (NMR)
- non frail (Other): No Fried's criteria
  Interventions: Diagnostic Test: Nuclear magnetic resonance (NMR)

INTERVENTIONS:
Diagnostic Test: Nuclear magnetic resonance (NMR) — Muscle architecture, lipid and active tissue muscle content should be measured. Proton NMR imaging (MRI)

SUMMARY:
Frailty is a multideterminant syndrome in which muscle function appears to play a central role. Muscle function depends on brain control, nutrition and perfusion. We hypothesized that multiparametric MRI assessment combined with comprehensive gerontological assessment (CGA) and routine biological assessment of inflammation in a sample of older people with and without diabetes will allow to explore on one side the possibilities of multi-parametric MRI muscle and brain imaging to describe the correlates of frailty and on the other side will describe the different muscle/brain alterations due to diabetes in frailty.

The main objective is to compare the lipid percent of the rectus femoris in frail and pre-frail older subjects and in non-frail older subjects.

DETAILED DESCRIPTION:
Frailty concept has been created to screen the older people at risk for dependency and to propose preventive intervention. Muscle function is at the centre of the concept and the majority of interventions proposed to reverse or to prevent frailty have targeted physical function. Anatomical and functional alteration of muscle, called sarcopenia is defined as a low skeletal muscle mass, a decrease in strength (dynapenia or sarcopenia is the age-associated loss of muscle strength that is not caused by neurologic or muscular diseases) and functional consequences such as low gait speed. Qualitative analysis should be associated with quantitative (mass) analysis in older subjects assessed for frailty. Muscle architecture, lipid and active tissue muscle content should be measured. Proton NMR imaging (MRI) can be used for this purpose. Brain changes were also reported to be associated with frailty. The study of structural changes associated with brain MRI alterations may better explain the frailty process.

Robust, frail and pre-frail subjects will be compared for clinical and MRI data. Grey matter volumes, white matter hyperintensities, diffusion tensor imaging data and muscle assessments relationships will be described After baseline assessment follow-up will be performed by phone calls after one month and after six months to record the number of falls and severity, the number of unscheduled hospitalization, the admission in institution for older people and death.

ELIGIBILITY:
Inclusion Criteria:

* Robust or frail or pre-frail with at least 25% frail and 25% pre-frail according to Frieds criteria
* Barthel index > or = 60/100
* With or without diabetes mellitus, 45 to 55 % with known diabetes mellitus
* With no contraindication to undergo an MRI examination

Exclusion Criteria:

* not willing to participate
* not able to give informed consent or to understand basic instruction due to any problem (sensorial, educational, language)
* without social insurance
* with a legal protection
* with significant cognitive alteration (MMSe<21/30 or in case of low literacy <19/30)
* with a recent (2 month period) severe event: hospitalization, sepsis, stroke even with complete recovery, trauma
* with stroke sequelae (motor, speech)

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-18 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Fat involution and trophicity in rectus femoris | day 1
  percentage of the rectus femoris lipid of both leg (dominant and non-dominant) in frail and pre-frail older subject and in non-frail older subjects (MRI with T1)

SECONDARY OUTCOMES:
description of brain by MRI | day 1
  description of MRI brain correlates of frailty and assessment of their sensibility / specificity with regards to Fried's frailty syndrome in a population older than 70y with at least 25% of subjects frail and 25% pre-frail and none with high level of daily living dependency.
Evaluation of inflammation grade | day 1
  description of muscle/brain MRI correlates of frailty and assessment of their sensibility / specificity with regards to Fried's frailty syndrome in a population with low/medium grade inflammation (HsCRP>3mg/L), older than 70y as compared to other subjects
measure the myostatin rate | day 1
  To explore the role of Myostatin in the regulation loop of muscle function during frailty
measure the cystatin-C and creatinine rate | day 1
  Determine the associations between muscle alterations seen on MRI and glomerular filtration rate estimated using serum cystatin-C or creatinine
measure the serum interleukin IL-1b and IL-18 rate | day 1
  Determine the associations between muscle alterations seen on MRI and serum IL-1b and IL-18.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle BOURDEL-MARCHASSON, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - Service de Médecine Gériatrique, CHU de LIMOGES, Limoges
  - Service de gériatrie - CHU Bordeaux - hôpital Xavier Arnozan, Pessac

IPD SHARING:
Plan to Share IPD: No